CLINICAL TRIAL: NCT07291050
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of TQB3217 Tablets in Subjects With Advanced Malignant Tumors
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of TQB3217 Tablets in Subjects With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3217-I-01
Record Dates: First submitted 2025-12-07; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3217Tablets (Experimental): TQB3217 Tablets: Administer once daily, recommended to be taken orally on an empty stomach in the morning at a fixed time, continuously, with each 21-day period as one treatment cycle.
  Interventions: Drug: TQB3217Tablets

INTERVENTIONS:
Drug: TQB3217Tablets — TQB3217 Tablets are ubiquitin specific peptidase 1(USP1)-t inhibitor.

SUMMARY:
This is the first-in-human clinical study of TQB3217, aiming to evaluate the safety, tolerability, and pharmacokinetic characteristics of TQB3217 in advanced solid tumors, and to preliminarily explore its efficacy in solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* Gender is not restricted; Age: 18 to 75 years old; an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; expected survival period ≥ 3 months;
* Patients with histologically or cytologically confirmed advanced malignant solid tumors that have failed standard treatment (disease progression or intolerance) or for which there is no standard treatment plan;
* The main organs function well;
* Women of childbearing age should take effective contraceptive measures during the study and within 6 months after the end of the study; serum or urine pregnancy test must be negative within 7 days before enrollment, and they must be non-lactating subjects; men must agree to take effective contraceptive measures during the study and within 6 months after the end of the study.

Exclusion Criteria:

* History of other malignant tumors within 3 years prior to the first administration of the study drug;
* Has multiple factors affecting oral medication;
* Unalleviated toxicity ≥ grade 1 above CTCAE v5.0 due to any previous therapy, excluding hair loss;
* Major surgical treatment, open biopsy and obvious traumatic injury were performed within 28 days before the study, or have not fully recovered from previous surgery, or are expected to require major surgical surgery during the study period;
* Arteriovenous thrombotic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism;
* Patients who have epilepsy and need treatment or have a history of epileptic seizures, consciousness disorders or unexplained coma within the last 12 months;
* Have a history of psychotropic drug abuse and can not quit or have mental disorders;
* Subjects with any severe and / or uncontrolled disease;
* Has known symptomatic central nervous system metastases and/or cancerous meningitis;
* Presence of massive serous pleural/abdominal/pericardial effusion with clinical symptoms or requiring repeated drainage.
* Has participated in other clinical trials within 4 weeks before first dose;
* Receipt of chemotherapy or immunotherapy within 4 weeks before the first administration;, Receipt of radiotherapy or small molecule targeted drugs within 2 weeks, or are still within 5 half-lives of the drugs;
* Receipt of Chinese patent medicines explicitly indicated for anti-tumor use in their drug labels approved by National Medical Products Administration (NMPA) within 2 weeks prior to the first administration;
* According to the judgement of the investigators, Subjects who are at risk of active bleeding during the trial period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 days)
  DLT refers to occurrence of drug-related adverse events within the first treatment cycle after subjects receive single-dose or multiple-dose treatment, as defined by the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 toxicity assessment criteria.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 21 days)
  MTD is defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended Phase II Dose (RP2D) | Baseline up to 24 months
  DLT describes side effects of a drug or other treatment that are serious enough to evaluate RP2D of TQB3217 tablets in adult patients with advanced malignant cancer.

SECONDARY OUTCOMES:
Numbers of participant with Adverse events (AEs) and serious adverse events (SAEs) | 30 days after the last administration
  The incidence and severity of AEs and SAEs, as well as abnormal laboratory test indicators.
Time to Reach the Maximum Plasma Concentration (Tmax) | Single dose day 1: pre-dose, at 0.5, 1, 1.5，2, 3, 4, 6, 8, 12, 24, 48, 72 hours post dose. Days 7, 14 and 21 of multiple dosing cycle 1: pre-dose. Day 21 of multiple dosing cycle 1: at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose (21 days a cycle)
  To characterize the pharmacokinetics of TQB3217 by assessment of time to reach maximum plasma concentration after single and multiple dosing.
Peak concentration (Cmax) | Single dose day 1: pre-dose, at 0.5, 1, 1.5，2, 3, 4, 6, 8, 12, 24, 48, 72 hours post dose. Days 7, 14 and 21 of multiple dosing cycle 1: pre-dose. Day 21 of multiple dosing cycle 1: at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose (21 days a cycle)
  The maximum observed plasma concentration of TQB3217 tablets.
Half-life (t1/2) | Single dose day 1: pre-dose, at 0.5, 1, 1.5，2, 3, 4, 6, 8, 12, 24, 48, 72 hours post dose. Days 7, 14 and 21 of multiple dosing cycle 1: pre-dose. Day 21 of multiple dosing cycle 1: at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose (21 days a cycle)
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Area under the concentration-time curve (AUC [0-infinity] | Single dose day 1: pre-dose, at 0.5, 1, 1.5，2, 3, 4, 6, 8, 12, 24, 48, 72 hours post dose. Days 7, 14 and 21 of multiple dosing cycle 1: pre-dose. Day 21 of multiple dosing cycle 1: at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose (21 days a cycle)
  To characterize the pharmacokinetics of TQB3217 by assessment of area under the plasma concentration time curve from 0 extrapolated to infinity.
Area under the concentration-time curve (AUC [0-t] | Single dose day 1: pre-dose, at 0.5, 1, 1.5，2, 3, 4, 6, 8, 12, 24, 48, 72 hours post dose. Days 7, 14 and 21 of multiple dosing cycle 1: pre-dose. Day 21 of multiple dosing cycle 1: at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose (21 days a cycle)
  To characterize the pharmacokinetics of TQB3217 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Apparent clearance (CL/F) | Single dose day 1: pre-dose, at 0.5, 1, 1.5，2, 3, 4, 6, 8, 12, 24, 48, 72 hours post dose. Days 7, 14 and 21 of multiple dosing cycle 1: pre-dose. Day 21 of multiple dosing cycle 1: at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose (21 days a cycle)
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Apparent Volume of Distribution during the Terminal Phase | Single dose day 1: pre-dose, at 0.5, 1, 1.5，2, 3, 4, 6, 8, 12, 24, 48, 72 hours post dose. Days 7, 14 and 21 of multiple dosing cycle 1: pre-dose. Day 21 of multiple dosing cycle 1: at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose (21 days a cycle)
  Apparent volume of distribution during the Terminal Phase of the TQB3217 in plasma.
Objective Response Rate (ORR) | Up to 2 years
  The percentage of complete response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.
Disease control rate (DCR) | Up to 2 years
  Defined as the proportion of subjects with Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
Duration of Response (DOR) | Up to 2 years
  Defined as the time from first documented response to documented disease progression.
Overall Survival (OS) | From start of study treatment up to die ，estimated at two years
  the time from start of study treatment to date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China